CLINICAL TRIAL: NCT01556152
Title: A Phase II, 4 Week Randomized, Double-Blind, Parallel Group, Placebo Controlled Proof of Concept Study to Evaluate Efficacy, Safety and Tolerability of GRC 17536 in Patients With Painful Diabetic Neuropathy
Brief Title: A Clinical Trial to Study the Effects of GRC 17536 in Patients With Painful Diabetic Neuropathy (Painful Extremities Due to Peripheral Nerve Damage in Diabetic Patients)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to new scientific evidence assessment, the study design was revised before the study started recruitment
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRC 17536-201; 2011-005879-16 (EudraCT Number)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Arm 1 (Active Comparator)
  Interventions: Drug: GRC 17536 (Medium Dose)
- Traetment Arm 2 (Active Comparator)
  Interventions: Drug: GRC 17536 (Low Dose)
- Treatment Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRC 17536 (Medium Dose) — 1 BD for 28 days
  Arms: Treatment Arm 1
Drug: GRC 17536 (Low Dose) — 1 BD for 28 Days
  Arms: Traetment Arm 2
Drug: Placebo — Matching Placebo for 28 Days
  Arms: Treatment Arm 3

SUMMARY:
Diabetic peripheral neuropathy (DPN) represents a diffuse symmetric and length-dependent injury to peripheral nerves that has major implications on quality of life (QOL), morbidity, and costs from a public health perspective. Painful diabetic neuropathy affects 16% of patients with diabetes. Pharmacological agents used in the management of painful DPN mainly include tricyclic antidepressants, selective serotonin and norepinephrine reuptake inhibitors, opioids, and anti epileptic drugs. However, only two drugs (duloxetine and pregabalin) have been formally approved by the EMEA and the US FDA for the treatment of painful DPN. Generally, the available treatment options do not give total relief, are not effective in all patients, and only about one-third of patients may achieve more than 50% pain relief. Hence newer therapies are required for the treatment of DPN.

This is randomized, double-blind, placebo-controlled, parallel group study. The study will include patients with type 1 or type 2 diabetes mellitus with history of pain attributed to DPN for least 6 months and no greater than 5 years.

Patients will be recruited after providing written informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to provide voluntary written informed consent
2. Male and female (women of non child-bearing potential) patients ≥18 yrs and ≤ 75 yrs
3. Patients with diabetes mellitus with painful peripheral neuropathy for at least 6 months
4. A baseline 24-hour average daily pain intensity score ≥5
5. Women must be of non child-bearing potential, defined as post menopausal or surgically sterile.

Exclusion Criteria:

1. Other chronic pain conditions not associated with DPN, that may confound the assessment of neuropathic pain
2. Other causes of neuropathy or lower extremity pain
3. Complex regional pain syndrome or trigeminal neuralgia
4. Lower extremity amputations other than toes
5. Participation in another study with an investigational compound within the previous 90 days prior to study medication administration, or concurrent participation in another clinical study
6. Major depression.
7. Presence or history of cancer within the past 5 years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.
8. Patients with clinically significant or uncontrolled hepatic, gastrointestinal, cardiovascular, respiratory, neurological (other than neuropathy), psychiatric, hematological, renal, or dermatological disease, or any other medical condition that according to Investigator's medical judgment: Could interfere with the accurate assessment of safety or efficacy, or, Could potentially affect a patient's safety or study outcome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour average pain intensity (API) score | 4 weeks

SECONDARY OUTCOMES:
Mean night-time API Score | 4 weeks
Patient Global Impression of Change | 4 weeks
Clinician Global Impression of Change | 4 weeks
Adverse events (AE) | 4 weeks
Pharmacokinetics: Cmax, Tmax, AUC 0-tau, AUC0-24 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kavita Muchandi, MD, Study Director — Glenmark Pharmaceuticals Ltd
Locations (2):
- Site 2, Mainz, Germany
- Site 1, Manchester, United Kingdom